CLINICAL TRIAL: NCT01022710
Title: Early Detection of Noise-Induced Hearing Loss
Status: Withdrawn | Type: Observational
Why Stopped: We did not enroll any subjects because we realized we needed to establish the technique more definitively before proceeding to human testing.
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: C7107-R; 00860 (Other Grant/Funding Number: Department of Veterans Affairs)
Record Dates: First submitted 2009-11-25; First posted 2009-12-01 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Hearing Loss, Sensorineural
Keywords: hearing loss; otoacoustic emissions
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — No biospecimens will be collected for this study
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Veterans with sensorineural hearing loss

SUMMARY:
This study measures sounds produced by the sensory receptors of the inner ear called hair cells. These sounds are called otoacoustic emissions and one special case the investigators are studying are called distortion product otoacoustic emissions (DPOAEs) produced by presenting two tones to the ear. If the ear is damaged by noise exposure DPOAEs are reduced. In this study the investigators are attempting to improve the DPOAE test by adding a third tone to make the test more frequency specific. Whether the third tone helps will be determined by comparing DPOAEs collected with and without the third tone to clinical audiograms. If the addition of the third tone helps then the investigators expect DPOAEs tracked as a function of frequency (DP-grams) will more closely match the clinical audiograms.

DETAILED DESCRIPTION:
The overall goal of the proposed research is to identify features of distortion product otoacoustic emissions (DPOAEs) that will eventually improve clinical methods for the early detection of noise-induced hearing loss (NIHL), which is a major sensory disability suffered by military Veterans, in particular. Toward this end, a special-purpose DPOAE measure the investigators call an augmented will be obtained. These DP-grams will test the notion that subtle post-noise changes in the DPOAE response space can be more sensitively identified when the f2 and basal source DPOAEs are isolated by the use of an interference tone (IT) and vector subtraction methods than by the commonly employed standard DP-gram procedures. The term 'augmented' maps or DP-grams was coined to describe these frequency functions when obtained with the IT present in that, under this condition, the basal source that 'fills in' or 'masks' the damage pattern is removed. The discovery of the contaminating basal source promises to modify the hearing field's current knowledge concerning the fundamental processes underlying DPOAE generation, and may also lead to the development of DPOAE tests that more sensitively identify the earliest stages of NIHL. Such tests may also be useful in Veterans, who are clinic patients and often have significant preexisting hearing losses in that higher-level primary tones can be used to increase the signal-to-noise ratio (SNR) while maintaining their sensitivity and frequency specificity. The investigators will test the ability of augmented DP-grams elicited by higher-level primary tones to uncover damaged regions in Veterans with NIHL. The notion examined here is that high-level primary tones will be more useful under conditions of preexisting hearing loss than conventional low-level primaries using the optimized augmented DP-gram by removing basal sources that come into play to obscure damaged cochlear regions as primary-tone levels are increased. Together, the combined experiments will provide a more complete understanding of the generation of DPOAEs, which will permit the creation of a useful clinical test for diagnosing and monitoring the development of NIHL.

ELIGIBILITY:
Inclusion Criteria:

* Veterans 18-65 years old

Exclusion Criteria:

* Individuals with no measurable distortion-product otoacoustic emissions (DPOAEs) since the goal of the study is to relate DPOAEs to hearing function

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Veterans reporting to the VA Loma Linda Healthcare System identified with sensorineural hearing loss
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
DP-gram with interference tone 1/3 octave above f2 | At the end of the testing session

CONTACTS AND LOCATIONS:
Overall Officials: Glen K Martin, PhD, Principal Investigator — VA Loma Linda Healthcare System, Loma Linda, CA
Locations (1):
- VA Loma Linda Healthcare System, Loma Linda, CA, Loma Linda, California, United States

REFERENCES:
- [Result] Martin GK, Stagner BB, Fahey PF, Lonsbury-Martin BL. Steep and shallow phase gradient distortion product otoacoustic emissions arising basal to the primary tones. J Acoust Soc Am. 2009 Mar;125(3):EL85-92. doi: 10.1121/1.3073734. PMID 19275280
- [Result] Martin GK, Stagner BB, Lonsbury-Martin BL. Evidence for basal distortion-product otoacoustic emission components. J Acoust Soc Am. 2010 May;127(5):2955-72. doi: 10.1121/1.3353121. PMID 21117746
- [Result] Martin GK, Stagner BB, Chung YS, Lonsbury-Martin BL. Characterizing distortion-product otoacoustic emission components across four species. J Acoust Soc Am. 2011 May;129(5):3090-103. doi: 10.1121/1.3560123. PMID 21568412
- [Result] Martin GK, Stagner BB, Lonsbury-Martin BL. Time-domain demonstration of distributed distortion-product otoacoustic emission components. J Acoust Soc Am. 2013 Jul;134(1):342-55. doi: 10.1121/1.4809676. PMID 23862812